CLINICAL TRIAL: NCT03946540
Title: Follow up of Young People Treated in CAEDS 2009-2014. Longitudinal Follow Up of Eating Disorder Treatment
Brief Title: Longitudinal Follow Up of Eating Disorder Treatment
Acronym: L-FED
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Catherine Stewart, Senior Clinical Psychologist, South London and Maudsley NHS Foundation Trust
Other Study IDs: L-FED2019
Record Dates: First submitted 2019-04-10; First posted 2019-05-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Feeding and Eating Disorders of Childhood; Anorexia Nervosa; Bulimia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- L-FED sample: All young people treated in Maudsley Child and Adolescent Eating Disorder Service between 1/8/2009 and 31/1/2014.

SUMMARY:
The research proposed here seeks to delineate the outcomes of people who have received treatment for an eating disorder at a specialist eating disorder service in childhood or adolescence (hereafter 'former patients'). This will inform our understanding of the maintenance of treatment effects beyond initial trial follow-ups, and together with data collected during treatment will allow for identification of factors predicting chronicity which will inform further treatment development.

DETAILED DESCRIPTION:
Research Questions

1. Is recovery from an eating disorder in adolescence maintained and associated with good socio-economic outcomes?
2. Is poor outcome from eating disorder treatment in adolescence associated with a chronic course of illness?
3. Are there factors measured during treatment that predict maintenance of outcome or relapse?

This study will use a longitudinal follow up design, contacting former patients of the National and Specialist Child and Adolescent Mental Health Service (CAMHS) Eating Disorder Service, South London and Maudsley National Health Service (NHS) Foundation Trust (CAEDS) between 1/8/2009 and 31/1/2014. These former patients are now aged 16-27. The study will thus provide the longest and largest follow up of treated adolescents to date (n = 358 over a 4-8 year follow up). Former patients will be asked a series of questions by phone/post/email about their health and socio-economic well-being since discharge from the service. This data will be analysed together with assessment and outcome data collected while they were patients of CAEDS.

Measures Data will be collected using a data collection tool developed for this project, as well as the Eating Disorders Examination Questionnaire and the Work and Social Adjustment Scale.

Data collected will comprise:

* Age now
* Employment/education
* Any help sought for eating disorder
* Any help sought for other mental health difficulties
* Current weight
* Current binge/purge symptoms
* Current general well being All data will be self-reported by participants.

Statistical power The primary analysis will be descriptive. We will recruit as many of our original treatment group as possible.

A secondary analysis will be to predict who continues to require mental health care following discharge from CAEDS. Power has been calculated following Babyak's (2004) advice for power calculation for logistic regression of 13 events (continuing mental health care needs) per variable. We have taken figures from the original audit in which 24.1% (n = 69.89) had a poor outcome to hypothesise that a similar proportion of the sample at follow up will have a poor outcome. This is a conservative estimate given the chronicity of eating disorders in adulthood and the longitudinal data of on-going mental health difficulties even in the absence of diagnosable eating disorders. In order to run a logistic regression with 5 predictor variables will require 65 cases with on-going eating disorder symptoms. This will require recruitment of the majority of the original sample assuming the % of on-going difficulties remains the same. Depending on recruitment rate we will adjust analysis accordingly, and reduce the number of predictors in the model.

Data analysis

Planned analyses:

1. Descriptive analysis of key health and socio-economic outcomes for all young people who received treatment in the audited timeframe and split by treatment outcome and diagnosis for between group analysis.
2. Regression analysis to identify predictors of long term outcome from clinical variables measured at baseline assessment and service discharge (including weight, mood, anxiety, eating disorder symptoms)

ELIGIBILITY:
Inclusion criteria:

* People who were assessed and offered treatment at the National and Specialist CAMHS Eating Disorder Service, South London and Maudsley NHS Foundation Trust between 1/8/2009 and 31/1/2014.

Exclusion criteria:

* young people who were referred for treatment but did not attend assessment
* young people who were referred for treatment but did not meet criteria for an eating disorder
* young people who were referred for treatment but did not accept treatment (or attended for fewer than 3 sessions).

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People who were assessed and offered treatment at the National and Specialist CAMHS Eating Disorder Service, South London and Maudsley NHS Foundation Trust between 1/8/2009 and 31/1/2014
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2019-07-14 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Receipt of further treatment for an eating disorder in the first four years after discharge from treatment | From discharge from service to L-FED research assessment. Discharges between 2009 and 2014 (4-10) year follow up. Proportion of sample needing treatment in the first four years post discharge will be reported
  Self report of whether subsequent treatment for an eating disorder has been received since discharge. Self report of treatment received in the period between discharge and research follow up - including number and duration of outpatient treatment, hospital admission and day patient treatment. The four year outcome is the primary outcome as it allows for the most complete dataset for follow up.
Eating Disorder Examination Questionnaire (EDEQ). Fairburn & Beglin, 1994 | 28 days prior to L-FED research assessment
  Self reported eating disorder symptoms. This is a 28 item self report questionnaire which is scored using a 7 - point (0-6) rating scale. Four subscales are derived through adding together relevant items and diving by the number of items to give a score range for each subscale of 0-6. A total score is derived by adding together the subscales and diving by the number of subscales (ie 4) also giving a score range of 0-6. Higher scores indicate greater impairment.
Work and social adjustment scale (WSAS) Mundt, J. C., I. M. Marks, et al. (2002). | At time of L-FED research assessment. Discharges between 2009 and 2014 (4-10) year follow up. Variation in time since discharge will be stratified in analysis.
  Self reported impact of symptoms on functioning. This is a self report measure of the impact of illness on work and social functioning. It is a five item questionnaire with each item scored 0-8 giving a total score range of 0-40 where high scores indicate greater impairment.

SECONDARY OUTCOMES:
Receipt of treatment for an eating disorder >4 years after discharge from treatment | From four years post discharge from service to L-FED research assessment. Proportion
  Self report of whether subsequent treatment for an eating disorder has been received since discharge. Self report of treatment received in the period between discharge and research follow up - including number and duration of outpatient treatment, hospital admission and day patient treatment. >4 years post treatment is a secondary outcome because for some participants will not have been out of treatment for more that 5 years. We will report on the proportion of those who have been discharged for each time period who have required subsequent treatment (eg % of those discharged for 8+ years who have required further treatment)
Psychosocial wellbeing | At time of L-FED assessment.Discharges between 2009 and 2014 (4-10) year follow up. Variation in time since discharge will be stratified in analysis.
  Self report questionnaire assessing function and well-being. This is a study specific tool which measures education, employment, and subjective experience of well-being.

OTHER OUTCOMES:
Receipt of treatment for any other mental health difficulties in four years post discharge, and at >4 years post discharge. | 1: Up to four years post discharge. 2: as applicable up to 10 years post discharge as described able for receipt of treatment for an eating disorder
  Self report of receipt of treatment for other mental health difficulties since discharge
Self harm since discharge | Four time points assesed: while in treatment, since discharge, in the past three months on in the past month. Variation in time since discharge will be stratified in analysis.
  Self report of self harm while in treatment, since discharge, in the past three months and in the past month.
Current eating disorder symptoms | At time of L-FED assessment. Discharges between 2009 and 2014 (4-10) year follow up. Variation in time since discharge will be stratified in analysis.
  Study specific questions assessing whether others consider weight to be in a healthy range, express concerns about eating, menstruation (where applicable) and current weight and height.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine s Stewart, }hD DClinPsy, Principal Investigator — South London and Maudsley NHS Foundation Trust
Locations (1):
- Maudsley Centre for Child and Adolescent Eating Disorders, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No